CLINICAL TRIAL: NCT05876351
Title: Prospective, Single-Arm, Multicenter Study to Evaluate the Efficacy, Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Eculizumab in Complement Inhibitor Treatment-Naïve Pediatric and Adult Participants With Atypical Hemolytic Uremic Syndrome (aHUS) in China
Brief Title: Eculizumab in Pediatric and Adult Participants With Atypical Hemolytic Uremic Syndrome (aHUS) in China
Acronym: Soliris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7413C00001; ECU-aHUS-302 (Other: Alexion); 2025-000162-29 (EudraCT Number)
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Atypical Hemolytic Uremic
Keywords: atypical hemolytic uremic; aHUS
MeSH Terms: interventions — eculizumab

STUDY DESIGN:
Intervention Model Description: open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eculizumab (Experimental): Participants will receive Eculizumab in a single dose vial.
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Weight-based doses of Eculizumab will be administered intravenously as an induction dose followed by maintenance dose at Day 8, 15, or 29 depending on weight; then every 2 or 3 weeks, depending upon weight.

SUMMARY:
This is a Phase 3b, open-label, single-arm, multicenter study to evaluate the efficacy and safety of eculizumab in participants with atypical hemolytic uremic syndrome (aHUS) in China

DETAILED DESCRIPTION:
This is a Phase 3b, open-label, single-arm, multicenter study to evaluate the efficacy and safety of eculizumab in participants with aHUS in China. The study will be conducted in participants of any age who weigh ≥ 5 kg and who previously have not been treated with complement inhibitors. The study consists of an up to 7-day Screening Period and a 26-week Treatment Period. An 8-week Safety Follow-up Phone Call will be required only for participants who discontinue eculizumab treatment during the study or for participants who will not receive continued access to eculizumab after completing study treatment. Approximately 25 eligible participants in China will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Any age weighing ≥ 5 kg
2. Complement treatment naïve with evidence of TMA.
3. History of aHUS prior to kidney transplant,or persistent evidence of TMA at least 4 days after modifying the immunosuppressive regimen.
4. Among participants with onset of TMA postpartum, persistent evidence of TMA for > 3 days after the day of childbirth
5. All participants must be vaccinated against N meningitidis if not already vaccinated within the time period of active coverage specified by the vaccine manufacturer.
6. Participants < 18 years of age must have been vaccinated against Haemophilus influenzae type b (Hib) and Streptococcus pneumoniae according to local vaccination schedule guidelines.
7. In participants receiving treatment with medications known to cause TMA, persistent evidence of TMA at least 4 days after modifying the excluded medication

Exclusion Criteria:

1. Known familial or acquired ADAMTS13deficiency (activity < 5%).
2. ST-HUS as demonstrated by local guidelines.
3. Positive direct Coombs test which is indicative of a clinically significant immune-mediated hemolysis not due to aHUS.
4. HIV infection, and /or unresolved meningococcal disease
5. Ongoing sepsis, and / or presence or suspicion of active and untreated systemic infection
6. Organ transplantation history, and/or Bone marrow transplant/hematopoietic stem cell transplant within 6 months prior to the start of Screening.
7. Among participants with a kidney transplant, acute kidney dysfunction within 4 weeks of transplant consistent with the diagnosis of acute antibody-mediated rejection.
8. Among participants without a kidney transplant, history of kidney disease other than aHUS
9. Identified drug exposure-related HUS, and / or HUS related to vitamin B12 deficiency and / or known genetic defects of cobalamin C metabolism.
10. History of malignancy within 5 years of Screening.
11. Known systemic sclerosis (scleroderma), systemic lupus erythematosus, or antiphospholipid antibody positivity or syndrome.
12. Chronic dialysis.
13. Prior use of complement inhibitors.
14. Use of tranexamic acid within 7 days prior to the start of Screening.
15. Other immunosuppressive therapies.
16. Receiving chronic intravenous immunoglobulin (IVIg) within 8 weeks prior to the start of Screening.
17. Received vasopressors or inotropes within 7 days prior to Screening.
18. Previously or currently treated with a complement inhibitor.
19. Has participated in another interventional treatment study or used any experimental therapy.
20. Hypersensitivity to any excipient in eculizumab.
21. Pregnant or breastfeeding.

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Qingdao
  - Research Site, Taiyuan
  - Research Site, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7413C00001&attachmentIdentifier=1484821e-7ae9-457c-81aa-263cc2c205e5&fileName=Synopsis_ECU-aHUS-302_CSR_body_V1.0_-_signed_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After providing informed consent/assent, participants were screened for eligibility for the study during the 7-day Screening Period.
Groups:
- Eculizumab: Participants received eculizumab as an intravenous (IV) infusion at a dose and schedule according to body weight for 26 weeks.
Period: Overall Study
Arm/Group | Eculizumab
Started | 25
Received at Least 1 Dose of Study Drug | 25
Completed | 22
Not Completed | 3
Not completed — Other than specified | 2
Not completed — Study specific discontinuation criteria | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: Included all participants who received at least 1 dose of study intervention and had at least 1 efficacy assessment post first dose.
Groups:
- Eculizumab: Participants received eculizumab as an IV infusion at a dose and schedule according to body weight for 26 weeks.
Arm/Group | Eculizumab
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.40 (15.95) [lower limit 15.95]
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0
  Preterm newborn infants (gestational age < 37 wks) | 0
  Newborns (0-27 days) | 0
  Infants and toddlers (28 days-23 months) | 2
  Children (2-11 years) | 7
  Adolescents (12-17 years) | 2
  Adults (18-64 years) | 14
  From 65-84 years | 0
  85 years and over | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 25
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Complete Thrombotic Microangiopathy (TMA) Response
Description: The criteria for complete TMA response were:
  1. Normalization of platelet count (defined as platelet count ≥ 150000/microliter (ul).
  2. Normalization of lactate dehydrogenase (LDH, defined as LDH ≤ upper limit of normal [ULN]).
  3. ≥ 25% improvement in serum creatinine from baseline.
Time Frame: Up to Week 26
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 25
percentage of participants | 64.0 (42.5) [42.5 to 82.0]

2. Secondary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment.
  A serious AE (SAE) was defined as any untoward medical occurrence that, at any dose:
  * resulted in death,
  * was life-threatening,
  * required inpatient hospitalization or prolongation of existing hospitalization,
  * resulted in persistent disability/incapacity,
  * was a congenital anomaly/birth defect, or
  * was an important medical event.
  A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Adverse Events' Section.
Time Frame: Up to Week 34
Population: Safety Set: Included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 25
Participants
  Any AE | 24
  Any SAE | 8

3. Secondary Outcome: Mean Serum Concentration of Eculizumab
Time Frame: Pre-dose and post-dose at Days 1, 8, 29, 85, and 141; Pre-dose at Day 183
Population: Pharmacokinetic (PK) Analysis Set: Included all participants who received at least 1 dose of study intervention and had evaluable pharmacokinetic data. 'Number Analyzed' = number of participants evaluable at specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (ug/mL)
Arm/Group | Eculizumab
Number analyzed (Participants) | 25
micrograms per milliliter (ug/mL)
  Day 1: Pre-dose | 4.690 (0.00)
  Day 1: Post-dose | 373.423 (47.59)
  Day 8: Pre-dose: number analyzed (Participants) | 24
  Day 8: Pre-dose | 153.190 (69.69)
  Day 8: Post-dose: number analyzed (Participants) | 24
  Day 8: Post-dose | 498.262 (41.18)
  Day 29: Pre-dose: number analyzed (Participants) | 21
  Day 29: Pre-dose | 353.726 (36.96)
  Day 29: Post-dose: number analyzed (Participants) | 21
  Day 29: Post-dose | 727.862 (32.22)
  Day 85: Pre-dose: number analyzed (Participants) | 21
  Day 85: Pre-dose | 360.070 (43.89)
  Day 85: Post-dose: number analyzed (Participants) | 21
  Day 85: Post-dose | 728.624 (42.04)
  Day 141: Pre-dose: number analyzed (Participants) | 21
  Day 141: Pre-dose | 433.737 (41.32)
  Day 141: Post-dose: number analyzed (Participants) | 21
  Day 141: Post-dose | 883.675 (38.74)
  Day 183: Pre-dose: number analyzed (Participants) | 21
  Day 183: Pre-dose | 434.739 (38.66)

4. Secondary Outcome: Change From Baseline in Serum Free Complement 5 (C5)
Time Frame: Baseline (Day 1 pre-dose) to Days 1, 8, 29, 85 and 141 (pre-dose and post-dose) and pre-dose at Day 183
Population: Pharmacodynamic (PD) Analysis Set: Included all participants who received at least 1 dose of study intervention and had evaluable PD data. 'Number Analyzed' = number of participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Eculizumab
Number analyzed (Participants) | 25
ug/mL
  Day 1: Post-dose | -79.8842 (17.5197)
  Day 8: Pre-dose: number analyzed (Participants) | 24
  Day 8: Pre-dose | -79.6539 (17.8589)
  Day 8: Post-dose: number analyzed (Participants) | 24
  Day 8: Post-dose | -79.6636 (17.8610)
  Day 29: Pre-dose: number analyzed (Participants) | 21
  Day 29: Pre-dose | -80.4277 (17.1241)
  Day 29: Post-dose: number analyzed (Participants) | 21
  Day 29: Post-dose | -80.4284 (17.1241)
  Day 85: Pre-dose: number analyzed (Participants) | 21
  Day 85: Pre-dose | -80.0632 (17.3489)
  Day 85: Post-dose: number analyzed (Participants) | 21
  Day 85: Post-dose | -80.0632 (17.3489)
  Day 141: Pre-dose: number analyzed (Participants) | 21
  Day 141: Pre-dose | -80.0625 (17.3485)
  Day 141: Post-dose: number analyzed (Participants) | 21
  Day 141: Post-dose | -80.0632 (17.3489)
  Day 183: Pre-dose: number analyzed (Participants) | 21
  Day 183: Pre-dose | -80.0632 (17.3489)

5. Secondary Outcome: Change From Baseline in Serum Total C5
Time Frame: Baseline (Day 1 pre-dose) to Days 1, 8, 29, 85 and 141 (pre-dose and post-dose) and pre-dose at Day 183
Population: PD Analysis Set: Included all participants who received at least 1 dose of study intervention and had evaluable PD data. 'Number Analyzed' = number of participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Eculizumab
Number analyzed (Participants) | 25
ug/mL
  Day 1: Post-dose | -12.0267 (6.1396)
  Day 8: Pre-dose: number analyzed (Participants) | 24
  Day 8: Pre-dose | 37.9293 (21.3162)
  Day 8: Post-dose: number analyzed (Participants) | 24
  Day 8: Post-dose | 40.2831 (23.0175)
  Day 29: Pre-dose: number analyzed (Participants) | 21
  Day 29: Pre-dose | 65.9100 (25.0734)
  Day 29: Post-dose: number analyzed (Participants) | 21
  Day 29: Post-dose | 64.4783 (22.7695)
  Day 85: Pre-dose: number analyzed (Participants) | 21
  Day 85: Pre-dose | 71.2418 (25.7350)
  Day 85: Post-dose: number analyzed (Participants) | 21
  Day 85: Post-dose | 66.5267 (26.7232)
  Day 141: Pre-dose: number analyzed (Participants) | 21
  Day 141: Pre-dose | 71.8284 (25.3689)
  Day 141: Post-dose: number analyzed (Participants) | 21
  Day 141: Post-dose | 67.0693 (23.1231)
  Day 183: Pre-dose: number analyzed (Participants) | 21
  Day 183: Pre-dose | 78.5497 (27.1158)

6. Secondary Outcome: Number of Participants With an Anti-drug Antibody (ADA) Response
Description: An ADA response was defined as a positive ADA sample at any time during the study.
Time Frame: Up to Week 26
Population: Safety Set: Included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 25
Participants | 0

7. Secondary Outcome: Time to Complete TMA Response
Description: Time to complete TMA response was defined as the time from first infusion to the first time point at which all criteria for complete TMA response was met.
  The criteria for complete TMA response were:
  1. Normalization of platelet count (defined as platelet count ≥ 150000/ul.
  2. Normalization of LDH, defined as LDH ≤ ULN).
  3. ≥ 25% improvement in serum creatinine from baseline.
  Participants who did not have a response were censored at the date of last visit or study discontinuation at the time when the analysis was performed.
Time Frame: Up to Week 26
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Eculizumab
Number analyzed (Participants) | 25
days | 75.0 [22.0 to NA] — Upper limit was not reached due to limited number of events.

8. Secondary Outcome: Proportion of Participants On or Off Dialysis at Each Timepoint
Description: Participants were considered as 'off' dialysis at a specific time point if they were dialysis free for more than 5 days prior to that time point. Participants were considered as 'on' dialysis at a specific time point if they were dialysis free to 5 days or less up prior to that time point.
Time Frame: Baseline and Days 22, 43, 71, 99, 113, 127, 155 and 183
Population: Full Analysis Set: Included all participants who received at least 1 dose of study intervention and had at least 1 efficacy assessment post first dose. 'Number Analyzed' = number of participants evaluable at specified timepoint.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 25
proportion of participants
  Baseline: On Dialysis | 0.440 [0.244 to 0.651]
  Baseline: Off Dialysis | 0.560 [0.349 to 0.756]
  Day 22: On Dialysis: number analyzed (Participants) | 23
  Day 22: On Dialysis | 0.261 [0.102 to 0.484]
  Day 22: Off Dialysis: number analyzed (Participants) | 23
  Day 22: Off Dialysis | 0.739 [0.516 to 0.898]
  Day 43: On Dialysis: number analyzed (Participants) | 17
  Day 43: On Dialysis | 0.235 [0.068 to 0.499]
  Day 43: Off Dialysis: number analyzed (Participants) | 17
  Day 43: Off Dialysis | 0.765 [0.501 to 0.932]
  Day 71: On Dialysis: number analyzed (Participants) | 19
  Day 71: On Dialysis | 0.211 [0.061 to 0.456]
  Day 71: Off Dialysis: number analyzed (Participants) | 19
  Day 71: Off Dialysis | 0.789 [0.544 to 0.939]
  Day 99: On Dialysis: number analyzed (Participants) | 17
  Day 99: On Dialysis | 0.176 [0.038 to 0.434]
  Day 99: Off Dialysis: number analyzed (Participants) | 17
  Day 99: Off Dialysis | 0.824 [0.566 to 0.962]
  Day 113: On Dialysis: number analyzed (Participants) | 18
  Day 113: On Dialysis | 0.167 [0.036 to 0.414]
  Day 113: Off Dialysis: number analyzed (Participants) | 18
  Day 113: Off Dialysis | 0.833 [0.586 to 0.964]
  Day 127: On Dialysis: number analyzed (Participants) | 18
  Day 127: On Dialysis | 0.111 [0.014 to 0.347]
  Day 127: Off Dialysis: number analyzed (Participants) | 18
  Day 127: Off Dialysis | 0.889 [0.653 to 0.986]
  Day 155: On Dialysis: number analyzed (Participants) | 18
  Day 155: On Dialysis | 0.167 [0.036 to 0.414]
  Day 155: Off Dialysis: number analyzed (Participants) | 18
  Day 155: Off Dialysis | 0.833 [0.586 to 0.964]
  Day 183: On Dialysis: number analyzed (Participants) | 18
  Day 183: On Dialysis | 0.167 [0.036 to 0.414]
  Day 183: Off Dialysis: number analyzed (Participants) | 18
  Day 183: Off Dialysis | 0.833 [0.586 to 0.964]

9. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Each Scheduled Visit
Description: Expressed in milliliters per minute per 1.73 square meters of body surface area.
Time Frame: Baseline, Days 22, 43, 71, 99, 113, 127, 155 and 183
Population: Full Analysis Set: Included all participants who received at least 1 dose of study intervention and had at least 1 efficacy assessment post first dose. 'Number Analyzed' = number of participants evaluable at the specific timepoint. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number Analyzed' = number of participants evaluable at the specific timepoint.
Measure: Mean (Standard Deviation); unit: mL/min/1.73^2
Arm/Group | Eculizumab
Number analyzed (Participants) | 22
mL/min/1.73^2
  Day 22 | 39.82 (50.83)
  Day 43: number analyzed (Participants) | 16
  Day 43 | 32.72 (44.75)
  Day 71: number analyzed (Participants) | 18
  Day 71 | 40.33 (47.38)
  Day 99: number analyzed (Participants) | 16
  Day 99 | 37.53 (47.17)
  Day 113: number analyzed (Participants) | 17
  Day 113 | 35.88 (45.38)
  Day 127: number analyzed (Participants) | 17
  Day 127 | 35.85 (48.01)
  Day 155: number analyzed (Participants) | 16
  Day 155 | 43.33 (49.32)
  Day 183: number analyzed (Participants) | 17
  Day 183 | 36.29 (44.21)

10. Secondary Outcome: Proportion of Participants With a Chronic Kidney Disease (CKD) Stage Shift Categorized as "Improved", "Stable", or "Worsened" at Each Scheduled Visit Compared to Baseline
Description: CKD stage was classified based on the National Kidney Foundation Chronic Kidney Disease Stage where Stage 5 represents the most severe disease and Stage 1 represents the least severe disease.
  "Improved" excluded participants with Stage 1 at baseline as there was no room for improvement. "Worsened" excludes participants with Stage 5 at baseline as there was no room to worsen.
Time Frame: Baseline to Days 22, 43, 71, 99, 113, 127, 155 and 183
Population: Full Analysis Set: Included all participants who received at least 1 dose of study intervention and had at least 1 efficacy assessment post first dose. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number Analyzed' = number of participants evaluable at specified timepoint.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 22
proportion of participants
  Day 22: Improved | 0.545 [0.322 to 0.756]
  Day 22: Stable | 0.455 [0.244 to 0.678]
  Day 22: Worsened: number analyzed (Participants) | 7
  Day 22: Worsened | 0 [0 to 0.410]
  Day 43: Improved: number analyzed (Participants) | 16
  Day 43: Improved | 0.688 [0.413 to 0.890]
  Day 43: Stable: number analyzed (Participants) | 16
  Day 43: Stable | 0.313 [0.110 to 0.587]
  Day 43: Worsened: number analyzed (Participants) | 4
  Day 43: Worsened | 0 [0 to 0.602]
  Day 71: Improved: number analyzed (Participants) | 18
  Day 71: Improved | 0.722 [0.465 to 0.903]
  Day 71: Stable: number analyzed (Participants) | 18
  Day 71: Stable | 0.278 [0.097 to 0.535]
  Day 71: Worsened: number analyzed (Participants) | 5
  Day 71: Worsened | 0 [0 to 0.522]
  Day 99: Improved: number analyzed (Participants) | 16
  Day 99: Improved | 0.750 [0.476 to 0.927]
  Day 99: Stable: number analyzed (Participants) | 16
  Day 99: Stable | 0.250 [0.073 to 0.524]
  Day 99: Worsened: number analyzed (Participants) | 5
  Day 99: Worsened | 0 [0 to 0.522]
  Day 113: Improved: number analyzed (Participants) | 17
  Day 113: Improved | 0.765 [0.501 to 0.932]
  Day 113: Stable: number analyzed (Participants) | 17
  Day 113: Stable | 0.235 [0.068 to 0.499]
  Day 113: Worsened: number analyzed (Participants) | 6
  Day 113: Worsened | 0 [0 to 0.459]
  Day 127: Improved: number analyzed (Participants) | 17
  Day 127: Improved | 0.765 [0.501 to 0.932]
  Day 127: Stable: number analyzed (Participants) | 17
  Day 127: Stable | 0.235 [0.068 to 0.499]
  Day 127: Worsened: number analyzed (Participants) | 6
  Day 127: Worsened | 0 [0 to 0.459]
  Day 155: Improved: number analyzed (Participants) | 16
  Day 155: Improved | 0.875 [0.617 to 0.984]
  Day 155: Stable: number analyzed (Participants) | 16
  Day 155: Stable | 0.125 [0.016 to 0.383]
  Day 155: Worsened: number analyzed (Participants) | 5
  Day 155: Worsened | 0 [0 to 0.522]
  Day 183: Improved: number analyzed (Participants) | 17
  Day 183: Improved | 0.824 [0.566 to 0.962]
  Day 183: Stable: number analyzed (Participants) | 17
  Day 183: Stable | 0.176 [0.038 to 0.434]
  Day 183: Worsened: number analyzed (Participants) | 5
  Day 183: Worsened | 0 [0 to 0.522]

11. Secondary Outcome: Change From Baseline in Platelets
Description: Platelet values obtained from the day of a blood transfusion of platelets through 3 days after the transfusion are excluded from all analysis.
Time Frame: Baseline, Days 22, 43, 71, 99, 113, 127, 155, and 183
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: 10^9 platelets/liter (L)
Arm/Group | Eculizumab
Number analyzed (Participants) | 23
10^9 platelets/liter (L)
  Day 22 | 76.5 (117.7)
  Day 43: number analyzed (Participants) | 16
  Day 43 | 65.5 (90.1)
  Day 71: number analyzed (Participants) | 19
  Day 71 | 71.3 (97.9)
  Day 99: number analyzed (Participants) | 16
  Day 99 | 79.4 (68.1)
  Day 113: number analyzed (Participants) | 16
  Day 113 | 60.1 (82.7)
  Day 127: number analyzed (Participants) | 17
  Day 127 | 61.8 (86.1)
  Day 155: number analyzed (Participants) | 18
  Day 155 | 76.8 (98.2)
  Day 183: number analyzed (Participants) | 18
  Day 183 | 80.3 (98.0)

12. Secondary Outcome: Change From Baseline in LDH
Time Frame: Baseline, Days 22, 43, 71, 99, 113, 127, 155, and 183
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: microkatal per liter (ukat/L)
Arm/Group | Eculizumab
Number analyzed (Participants) | 23
microkatal per liter (ukat/L)
  Day 22 | -9.445 (12.459)
  Day 43: number analyzed (Participants) | 17
  Day 43 | -6.147 (10.175)
  Day 71: number analyzed (Participants) | 19
  Day 71 | -7.083 (10.099)
  Day 99: number analyzed (Participants) | 17
  Day 99 | -5.861 (8.356)
  Day 113: number analyzed (Participants) | 18
  Day 113 | -5.769 (8.041)
  Day 127: number analyzed (Participants) | 18
  Day 127 | -5.444 (8.314)
  Day 155: number analyzed (Participants) | 17
  Day 155 | -5.848 (8.478)
  Day 183: number analyzed (Participants) | 18
  Day 183 | -5.680 (8.172)

13. Secondary Outcome: Change From Baseline in Hemoglobin
Description: Hemoglobin values obtained from the day of a blood transfusion of either whole blood or packed red blood cells through 7 days after the transfusion are excluded from all analysis.
Time Frame: Baseline, Days 22, 43, 71, 99, 113, 127, 155, and 183
Population: Full Analysis Set: Included all participants who received at least 1 dose of study intervention and had at least 1 efficacy assessment post first dose. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number Analyzed' = number of participants evaluable at the specific timepoint.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Eculizumab
Number analyzed (Participants) | 23
grams per liter (g/L)
  Day 22 | 17.0 (18.3)
  Day 43: number analyzed (Participants) | 16
  Day 43 | 25.7 (20.1)
  Day 71: number analyzed (Participants) | 19
  Day 71 | 30.5 (22.6)
  Day 99: number analyzed (Participants) | 17
  Day 99 | 30.3 (19.3)
  Day 113: number analyzed (Participants) | 18
  Day 113 | 29.8 (17.8)
  Day 127: number analyzed (Participants) | 18
  Day 127 | 25.2 (16.4)
  Day 155: number analyzed (Participants) | 18
  Day 155 | 30.5 (14.9)
  Day 183: number analyzed (Participants) | 18
  Day 183 | 36.2 (15.8)

ADVERSE EVENTS:
Time Frame: Up to Week 34
Description: Safety Set: Included all participants who received at least 1 dose of study intervention.
Arm/Group | Eculizumab
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 8/25
Other Adverse Events (participants affected / at risk) | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eculizumab (N=25)
Bacterial infection (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Rotavirus infection (Infections and infestations) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eculizumab (N=25)
Bronchitis (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 3 (4)
Influenza (Infections and infestations) | 2 (2)
Respiratory tract infection (Infections and infestations) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 5 (8)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 7 (9)
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5)
Hepatic function abnormal (Hepatobiliary disorders) | 4 (5)
Pyrexia (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT05876351/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT05876351/SAP_001.pdf